CLINICAL TRIAL: NCT03923998
Title: Assessing Efficacy of Neoadjuvant Chemoradiotherapy as a Treatment Plan for Patients With Stage IVa Oral Cancer.
Brief Title: Adjuvant ChemoRadiotherapy Prior to Surgery in Stage IVa Oral Cancers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Indrayani Hospital and Cancer Institute (Other)
Collaborators: Tata Capital Limited (Unknown); Grant Medical Foundation Ruby hall Clinic (Unknown)
Responsible Party: Principal Investigator, Dr. Sanjay Deshmukh, Surgical Oncologist, Indrayani Hospital and Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OIT415
Record Dates: First submitted 2019-04-17; First posted 2019-04-23 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Squamous Cell Carcinoma of Oral Cavity
Keywords: Oral neoplasms; Mouth neoplasms
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Mouth Neoplasms | interventions — Neoadjuvant Therapy; Plastic Surgery Procedures; Mandibular Osteotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant chemoradiotherapy followed by surgery (Experimental): Preoperative chemotherapy with concurrent radiotherapy followed by definitive surgery
  Interventions: Drug: Neoadjuvant chemotherapy; Radiation: Neoadjuvant radiotherapy; Procedure: Resection and reconstruction

INTERVENTIONS:
Drug: Neoadjuvant chemotherapy — Three weekly concurrent chemotherapy with cisplatin 100 mg /m2
  Other Names: NACT
Radiation: Neoadjuvant radiotherapy — Preoperative radiotherapy over 5 weeks- Dose 180-200cgys per day/ total 4500 cgys
  Other Names: NACTRT
Procedure: Resection and reconstruction — Resection and reconstruction of mandibular/maxillary segment with prefabricated fibular graft
  Other Names: Mandibulectomy/Maxillectomy and reconstruction by free fibula flap

SUMMARY:
Oral cancer is the single largest cancer in males in India. 90-95% cases of oral cancer are Squamous cell carcinomas and many of them present at late stages (T3 and above). Treatment of OSCC includes single modality surgery, radiotherapy, or combinations of these modalities with or without systemic therapy. For unresectable cases, radiotherapy and/or chemotherapy is the treatment modality. Efficacy of neoadjuvant chemoradiotherapy for resectable stage IV tumors (late stage) needs to be evaluated to assess its benefit before surgery.

DETAILED DESCRIPTION:
This study will assess the benefit of preoperative adjuvant chemoradiotherapy in patients with an Stage IVa oral squamous cell carcinoma (OSCC). The study population will consist of patients who have not been treated previously. Patients satisfying the inclusion-exclusion criteria will be included in the study after obtaining a valid, written and informed consent. After reviewing the histopathological report, the patients will be treated as per the study protocol. The patients will be under regular follow-up with 3 monthly intervals for a period of one year and 6 monthly period in the following years. At each follow-up, patients will be evaluated clinically for evidence of locoregional tumor recurrence. The locoregional recurrence-free survival will be calculated based on the difference between the date of inclusion and the date of biopsy-proven recurrence. We will also record the overall survival, parameters like trismus, osteonecrosis and xerostomia. Quality of life will be assessed at a regular interval of 1 year using the University of Washington Quality of Life Questionnaire (UW-QOL v.4)

Study protocol:

1. Preoperative radiotherapy over 5 weeks- Dose 180-200cgys per day/ total 4500 cgys
2. Three weekly concurrent chemotherapy with cisplatin 100 mg /m2
3. Initial surgery in leg for Prefabrication of fibula - 2 weeks after starting of radiotherapy treatment. Delay is required for planning of implant position in the fibula.
4. Definitive surgical procedure with reconstruction by prefabricated flap, 6 weeks post radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed stage IVa squamous cell carcinoma of the oral cavity.
2. Surgically resectable oral squamous carcinoma with invasion of mandible or maxilla.
3. Newly diagnosed or previously untreated squamous cell carcinoma of the oral cavity.

Exclusion Criteria:

1. Patients with distant metastases.
2. Patients with contraindication to radiotherapy.
3. Patients with vascular disorders or ischemic heart disease. -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-03-15 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Objective response rate | Upto 1 year
  This will be deduced from pathological response in terms of complete and partial response. Complete response is defined as no invasive and no in situ residuals present in the surgical specimen. Partial response defined as at least a 30% reduction in the size of the lesion in the surgical specimen.
Disease free survival | 2 years
  Disease-free survival will be calculated as the time interval (months) between primary treatment and the first recurrence (whether local, regional or distant).
Overall Survival | 2 years
  Overall Survival will be calculated as the time interval (months) between primary treatment and death.

SECONDARY OUTCOMES:
Quality of life assessment | 2 years
  Patient reported quality of life will be assessed at a regular interval of 1 year using the University of Washington Quality of Life Questionnaire (UW-QOL v.4). The minimum score is 0 which is indicative of worse outcome while 100 is the maximum score and indicative of better outcome. Various parameters including chewing, pain, swallowing, saliva, appearance etc. are included in the questionnaire. Average score for each parameter with standard deviation will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Deshmukh, MS, Principal Investigator — Indrayani Hospital and Cancer Institute
Locations (1):
- Indrayani hospital and cancer institute, Pune, Maharshtra, India

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data for all primary and secondary outcomes will be made available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be made available 4 months post completion of the study.
Access Criteria: The data will be made available on request. Requestors will need to sign a data access agreement to obtain the data.